CLINICAL TRIAL: NCT01612637
Title: Can Pelvic Floor Muscle Training Reduce my Prolapse? A Randomised Controlled Trial Comparing the Effect of Pelvic Floor Muscle Training and Lifestyle Advice on Pelvic Organ Prolapse
Brief Title: Can Pelvic Floor Muscle Training Reduce my Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-4-2011-072
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2014-07

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic organ prolapse; Pelvic floor muscle training; Prolapse symptoms; Pelvic organ prolapse quantification system; Ultrasonography; Predictors
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Group 1 will be individually examined and instructed in pelvic floor muscle training before the intervention starts by specialized physiotherapists. The examination includes a vaginal or an anal examination. The women attend six group sessions within 12 weeks containing structured information about POP and the possible affection of POP on quality of life, exercising and sexual relationship. The lifestyle advice contains information about life style changes that could improve POP symptoms, such as bladder and bowel habits, coughing, heavy lifting, eating habits and weight loss. The women will perform pelvic floor muscle training in the group and they will perform pelvic floor muscle training at home. The training will be individually planned according to the findings of the pelvic floor physiotherapist. The women in the intervention group fill in an exercise diary and also describe on a Visual Analog Scale if the training causes any bother.
  Interventions: Behavioral: Pelvic floor muscle training and lifestyle advice
- Group 2 (Active Comparator): Group 2 attend six group sessions within 12 weeks containing structured information about POP and the possible affection of POP on quality of life, exercising and sexual relationship. The lifestyle advice contains information about life style changes that could improve POP symptoms, such as bladder and bowel habits, coughing, heavy lifting, eating habits and weight loss
  Interventions: Behavioral: Lifestyle advice

INTERVENTIONS:
Behavioral: Pelvic floor muscle training and lifestyle advice — Group 1 will be individually examined and instructed in pelvic floor muscle training before the intervention starts by specialized physiotherapists. The examination includes a vaginal or an anal examination. The women attend six group sessions within 12 weeks containing structured information about POP and the possible affection of POP on quality of life, exercising and sexual relationship and information that could improve POP symptoms, such as bladder and bowel habits, coughing, heavy lifting, eating habits and weight loss. The women will perform pelvic floor muscle training in the group and perform pelvic floor muscle training at home. The training will be individually planned according to the findings of the pelvic floor physiotherapist. The women in the intervention group fill in an exercise diary and also describe on a Visual Analog Scale if the training causes any bother.
  Arms: Group 1
Behavioral: Lifestyle advice — Group 2 attend six group sessions within 12 weeks containing structured information about POP and the possible affection of POP on quality of life, exercising and sexual relationship. The lifestyle advice contains information about life style changes that could improve POP symptoms, such as bladder and bowel habits, coughing, heavy lifting, eating habits and weight loss
  Arms: Group 2

SUMMARY:
Purpose The aim of this study is to examine if a structured pelvic floor muscle training combined with lifestyle advice with can improve pelvic organ prolapse (POP) symptoms more than structured lifestyle advice programme alone.

Background Pelvic organ prolapse (POP) is a common condition among adult women and almost one in ten women experience symptoms caused by POP. The key symptom of POP is seeing or feeling a bulge in the vaginal opening but POP often gives other symptoms, such as pain, difficulty emptying the bladder or the bowel, incontinence and sexual problems such as dyspareunia.

A majority of women with POP will be offered reconstructive surgery but the risk of reoperations is substantial and surgery may cause new symptoms. In one out of four women surgery does not relieve symptoms and the women have been exposed to unnecessary risk of complications.

It is therefore important to evaluate the effect of conservative treatments for POP. New studies have shown that pelvic floor muscle training offered in combination with lifestyle advice has a significant on POP symptoms and objective measures of POP compared to a lifestyle advice leaflet alone.

No studies have compared the effect of a combined pelvic floor muscle training and lifestyle advice programme with a structured programme of lifestyle advice and hypothetically the structured lifestyle advice programme could have a substantial effect on its own. Our hypothesis is that the pelvic floor muscle training is a vital component of a conservative treatment for POP.

Methods In this single-blind randomised controlled study women with POP will randomised to either a programme of structured pelvic floor muscle training combined with lifestyle advice or a structured lifestyle advice programme alone. Both groups will receive the same lifestyle advices through six (separate) lectures within 12 weeks. The training group will be examined and individually instructed in pelvic floor muscle training before the intervention starts and they will, in continuation with their lifestyle lectures, perform pelvic floor muscle training as group training

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age female reporting bothersome symptoms of any type of POP
* Newly referred to the hospital clinic
* Prolapse ≥II POP-Q
* Understand and write Danish

Exclusion Criteria:

* Instruction in pelvic floor muscle training within the last two years
* Dementia
* Pregnancy or less than one year postnatal
* Disorders that can affect ability to participate in the intervention such as neurological or psychiatric disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2012-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Patient Global Index of Improvement scale (PGI-I) | three months after ended intervention

SECONDARY OUTCOMES:
Objective pelvic organ prolapse measured with the pelvic organ prolapse Quantification system (POP-Q) | before, right after, three and 12 months after the intervention has ended
Pelvic Floor Distress Inventory - short form 20 (PFDI-20) | right after, three months and 12 months after ended intervention
  Validated condition-specific questionnaire
Pelvic Floor Impact Questionnaire - short form 7 (PFIQ-7) | right after, three months and 12 months after ended intervention
  Validated condition-specific questionnaire
Background variables | At time of inclusion
  age, parity, BMI, working status as predictors of effect of the intervention
Size of levator hiatus and presence of levator ani avulsions examined through transperineal ultrasound | At time of inclusion
  as predictors of effect of the intervention
Cost-effectiveness | 12 months after ended intervention
  Need for further treatment and calculation of economic costs for both interventions compared to number of surgeries avoided will be evaluated
Patient Global Index of Improvement scale (PGI-I) | Right after ended intervention and 12 months after ended intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital at Herlev, Copenhagen, Denmark